CLINICAL TRIAL: NCT02898155
Title: Are Potentially Avoidable Hospitalizations a Good Measure of Access To Primary Care in France?
Brief Title: Potentially Avoidable Hospitalisation in France
Acronym: HPE-LR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9670
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; COPD; Diabetes
Keywords: Avoidable hospitalizations; primary care; geographicvariation
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: measure of access to primary care and of the Interface Between Primary ans Secondary Care

SUMMARY:
Potentially Avoidable Hospitalizations (Pah) Are Studied As An Indirect Measure Of Access To Primary Care And Of The Interface Between Primary And Secondary Care. A Previous Work Unveils Considerable Geographic Variation In The Rate Of Pah In France And Suggest That Primary Care Organization Might Play A Role In This Variation. However, A Limitation Of This Work Lies In The Lack Of Data On Actual Primary Care Utilization.

The Aim Of This Study Is To Analyze The Role Of Primary Care In The Variation Of Potentially Avoidable Hospitalizations At the Zip Code Level, In The French Region Languedoc-Roussillon-Midi-Pyrénées.

The investigator will implement An Ecological Approach In Which The Geographic Variation In The Rate Of Pah Is Analyzed In The French Region Lrmp, Year 2014. Age- And Sex-Adjusted Rate Of Pah By Zip Codes (N=612) Is Modeled Using A Spatial Regression Model.

ELIGIBILITY:
Inclusion criteria:

* year 2014
* LRMP region
* Hospital admission in any public or private hospital

Exclusion criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with at least one hospital admission in the LRMP region in 2014.
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Rate of potentially avoidable admissions | 24 months

SECONDARY OUTCOMES:
Standardized Rate of potentially avoidable admissions | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire MERCIER, MD, PhD, Study Director — University Hospital, Montpellier; Gregoire mercier, MD, PhD, Study Chair — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No